CLINICAL TRIAL: NCT00830674
Title: A Phase I, Double-blind, Randomized, Placebo-controlled, Single-dose, Dose-escalation Study of KRN23 in X-linked Hypophosphatemia
Brief Title: A Study of KRN23 in X-linked Hypophosphatemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KRN23-US-02
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: XLH
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KRN23 (Experimental): Single IV or SC administration on day 1
  Interventions: Drug: KRN23
- Placebo (Placebo Comparator): Single IV or SC administration on day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — single dose IV or SC administration
  Arms: Placebo
Drug: KRN23 — Single IV administration on day 1: 0.003, 0.01, 0.03, 0.1 and 0.3 mg/kg and Single SC administration on day 1: 0.1, 0.3, 0.6 and 1.0 mg/kg
  Arms: KRN23

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of KRN23 after a single intravenous (IV) and subcutaneous (SC) administration in XLH patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Clinical diagnosis of XLH
3. TmP/GFR is less than 2.0 mg/dL
4. GFR is 60 mL/min or above

Exclusion Criteria:

1. Have any sign of active infectious disease or have had an infection requiring treatment with antibiotics within three weeks prior to screening
2. History of known immunodeficiency
3. Lactating females, female patients who are pregnant or planning to become pregnant during the study
4. Use of a pharmacologic vitamin D metabolite or its analog, phosphate, calcimimetics, and ingestion of aluminum hydroxide antacids within 10 days prior to screening and dosing
5. Use of any supplement contained phosphate, calcium and/or vitamin D within 10 days prior to screening and dosing
6. Receipt of live (attenuated) vaccine within 3-months prior to screening
7. Have any condition which, in the opinion of the Investigator, could present a concern for either patient safety or difficulty with data interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 7 weeks after dosing (maximally 11 weeks)
  AEs, etc

SECONDARY OUTCOMES:
Effect to pharmacodynamic parameter | Up to 7 weeks after dosing (maximally 11 weeks)
  Change in Serum Phosphate

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O. Carpenter, M.D., Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale University School of Medicine, New Haven, Connecticut
  - General Clinical Research Center, Indiana University School of Medicine, Indianapolis, Indiana
  - Duke Clinical Research Unit, Durham, North Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Derived] Carpenter TO, Imel EA, Ruppe MD, Weber TJ, Klausner MA, Wooddell MM, Kawakami T, Ito T, Zhang X, Humphrey J, Insogna KL, Peacock M. Randomized trial of the anti-FGF23 antibody KRN23 in X-linked hypophosphatemia. J Clin Invest. 2014 Apr;124(4):1587-97. doi: 10.1172/JCI72829. Epub 2014 Feb 24. PMID 24569459
- See also: KRN23-INT-002 An Extension Study of KRN23 in Adults With X-Linked Hypophosphatemia — http://www.clinicaltrials.gov/ct2/show/NCT01340482?term=KRN23&rank=1